CLINICAL TRIAL: NCT03414749
Title: Assessment of Balance Changes After Extremity Manipulation Therapy
Brief Title: Extremity Manipulation Impact on Postural Sway Characteristics
Acronym: Balance1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Parker University (Other)
Collaborators: University of Miami (Other); Whittier University (Unknown); University of Houston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Parker17_001
Record Dates: First submitted 2018-01-22; First posted 2018-01-30 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Healthy
Keywords: Chiropractic; postural sway; manipulation

STUDY DESIGN:
Intervention Model Description: This study used a randomized, crossover experimental design over three days of testing.
Who Masked: Participant, Outcomes Assessor
Masking Description: Treatment was unknown to outcome assessors. Participant were unaware of what the treatment would be and how it may / may not impact the outcome.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lower Extremity First (LEF) (Experimental): The treatment was a non-specific long-axis distraction to the ankle, knee, and hip provided was at the discretion of the clinic doctor (over 25 years experience).
  Interventions: Procedure: Lower Extremity First (LEF)
- Upper Extremity First (UEF) (Experimental): The treatment was a non-specific long-axis distraction to the shoulder, elbow and wrist provided was at the discretion of the clinic doctor (over 25 years experience).
  Interventions: Procedure: Upper Extremity First (UEF)

INTERVENTIONS:
Procedure: Lower Extremity First (LEF) — The intervention for the LEF group was a non-specific long-axis distraction to the ankle, knee, and hip or shoulder, elbow and wrist provided was at the discretion of the clinic doctor (over 25 years experience).
  Arms: Lower Extremity First (LEF)
Procedure: Upper Extremity First (UEF) — The intervention for the UEF group was a non-specific long-axis distraction to the shoulder, elbow and wrist provided was at the discretion of the clinic doctor (over 25 years experience).
  Arms: Upper Extremity First (UEF)

SUMMARY:
This study will evaluate the multi-segmental postural sway after upper versus lower extremity manipulation.

DETAILED DESCRIPTION:
The focus of this study is to explore the effect of upper and lower extremity chiropractic adjustments (manipulation) as well as surface condition (hard surface vs rocker board) on multisegmental postural control as represented by postural sway. Using a rocker (tilt) board, the participant cannot stand still, but has to adjust posture continuously to maintain balance. Body sways are considered to be self-induced because the design of the rocker board creates a natural instability without any external perturbation. This task provides a self-driven sensorimotor condition in addition to amplifying the sway dynamics. Because the rocker board has only one degree of freedom of motion, anteroposterior and lateral sways were considered separately on the device.

The investigators had the following hypotheses.

Hypothesis 1: Lower extremity adjustments will lead to reduced postural sway magnitude compared to upper extremity adjustments.

Hypothesis 2: Lower extremity adjustments will reduce sway variability of the rocker board, trunk and head compared to upper extremity adjustments.

Hypothesis 3: Lower extremity adjustments will facilitate the organization of sway behavior as assessed by the chaotic structure of sway.

ELIGIBILITY:
Inclusion Criteria:

* student in Parker University's Doctor of Chiropractic program and patient at the Parker University Wellness Clinic;
* available to take part in the study for all 3 test days;
* willing to forgo all non-normal daily activities and chiropractic treatments during the test days;

Exclusion Criteria:

* pregnant;
* previous major injury involving the extremities;
* previous surgeries to an extremity joint; and
* known neurological or systemic diseases.

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2017-07-24 (Actual); Primary Completion 2017-08-09 (Actual); Study Completion 2017-08-09 (Actual)

PRIMARY OUTCOMES:
Postural Assessment | Post Treatment on Day 1
  Each participant was fitted with two Shimmer3 sensors (Shimmer Sensing, Dublin, Ireland) on their head (occiput) and low back (over S2 tubercle) (see Figure 2) with a third Shimmer3 sensor placed on the surface (ground or rocker board). Participants were asked to perform a series of four postural tasks with two surface conditions (floor or rocker board) and two variations of each (eyes open or closed, and AP or ML rocker board direction). The conditions were randomized (using REDCap) such that either both floor or both rocker board conditions were performed first, with the remainder performed second. The order of variation within the surface type was held consistent for all occasions; eyes open then eyes closed on the floor, and AP then ML rotation direction on the rocker board.
Postural Assessment | Pre Treatment on Day 2
  Each participant was fitted with two Shimmer3 sensors (Shimmer Sensing, Dublin, Ireland) on their head (occiput) and low back (over S2 tubercle) (see Figure 2) with a third Shimmer3 sensor placed on the surface (ground or rocker board). Participants were asked to perform a series of four postural tasks with two surface conditions (floor or rocker board) and two variations of each (eyes open or closed, and AP or ML rocker board direction). The conditions were randomized (using REDCap) such that either both floor or both rocker board conditions were performed first, with the remainder performed second. The order of variation within the surface type was held consistent for all occasions; eyes open then eyes closed on the floor, and AP then ML rotation direction on the rocker board.
Postural Assessment | Post Treatment on Day 2
  Each participant was fitted with two Shimmer3 sensors (Shimmer Sensing, Dublin, Ireland) on their head (occiput) and low back (over S2 tubercle) (see Figure 2) with a third Shimmer3 sensor placed on the surface (ground or rocker board). Participants were asked to perform a series of four postural tasks with two surface conditions (floor or rocker board) and two variations of each (eyes open or closed, and AP or ML rocker board direction). The conditions were randomized (using REDCap) such that either both floor or both rocker board conditions were performed first, with the remainder performed second. The order of variation within the surface type was held consistent for all occasions; eyes open then eyes closed on the floor, and AP then ML rotation direction on the rocker board.
Postural Assessment | Pre Treatment on Day 3
  Each participant was fitted with two Shimmer3 sensors (Shimmer Sensing, Dublin, Ireland) on their head (occiput) and low back (over S2 tubercle) (see Figure 2) with a third Shimmer3 sensor placed on the surface (ground or rocker board). Participants were asked to perform a series of four postural tasks with two surface conditions (floor or rocker board) and two variations of each (eyes open or closed, and AP or ML rocker board direction). The conditions were randomized (using REDCap) such that either both floor or both rocker board conditions were performed first, with the remainder performed second. The order of variation within the surface type was held consistent for all occasions; eyes open then eyes closed on the floor, and AP then ML rotation direction on the rocker board.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine A Pohlman, DC, MS, Study Director — Parker University
Locations (1):
- Parker University, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make IPD available.